CLINICAL TRIAL: NCT02917759
Title: Establishment of a Tissue and Blood Registry to Support Translational Investigations Into the Biology, Etiology and Therapy of Liver and Biliary Tumors
Brief Title: Liver and Biliary Tumor Tissue Registry
Status: Terminated | Type: Observational
Why Stopped: Lack of funding to support enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tushar Patel, Consultant, Mayo Clinic
Other Study IDs: 13-006829
Record Dates: First submitted 2016-09-24; First posted 2016-09-28 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma; Cholangiocarcinoma
Keywords: liver cancer; biliary tract cancer; cholangiocarcinoma; hepatocellular carcinoma; liver tumor; biliary tumor; hepatoma; liver mass
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Liver Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — whole blood and tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hepatocellular cancer: Surgical waste tissue will be collected after removal of a liver tumor. A blood sample may be collected at the time of labs related to treatment for the diagnosis. An extra sample of biopsy tissue will be collected from participants having a targeted mass biopsy.
- Cholangiocarcinoma: Surgical waste tissue will be collected after removal of a biliary tumor. A blood sample may be collected at the time of labs related to treatment for the diagnosis. An extra sample of biopsy tissue will be collected from participants having a targeted mass biopsy.

SUMMARY:
Patients having surgery to remove a liver or biliary tissue mass or having a biopsy of a mass or lesion will have a tissue sample collected and stored for future research of liver and biliary diseases. A blood sample may also be collected at the time of enrollment.

DETAILED DESCRIPTION:
The study establishes a tissue and blood registry at Mayo Clinic Florida to support translational investigations into the biology, etiology and prognosis of liver and biliary masses such as through the use of patient-derived xenografts.

Patients having surgery to remove a liver or biliary mass or having a biopsy of a mass or lesion will be asked to donate a portion of the removed mass for research purposes. Only portions of the mass not required for clinical diagnostic evaluation, or surgical waste, will be used in this research study.

The tissues acquired will be stored and used for any specific, hypothesis driven protocols that are IRB approved. Serum and plasma samples may also be obtained at enrollment.

Clinical patient data from medical charts that may be correlative to outcomes will be collected and stored in a password secure data base. Data will be extracted from medical records charts.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo surgical resection of a liver or biliary mass

Exclusion Criteria:

* Under 18 years of age. Prior radiation to mass.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals undergoing surgical removal of a liver or biliary mass at Mayo Clinic Florida
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-02; Primary Completion 2025-12 (Actual); Study Completion 2025-12 (Actual)

PRIMARY OUTCOMES:
Number of successful xenografts established | 6 months
  The number of successful individual patient derived xenografts that are established beyond the second passage in immunodeficient mice

CONTACTS AND LOCATIONS:
Overall Officials: Tushar C Patel, MBChB, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials